CLINICAL TRIAL: NCT03910920
Title: Cross Transmissions of Pseudomonas Aeruginosa in a Pediatric Cohort Followed-up at the Cystic Fibrosis Reference Center of the Queen Fabiola Children's University Hospital.
Brief Title: Cross Transmissions of Pseudomonas Aeruginosa Between Children From a Same Cystic Fibrosis Center.
Acronym: PAPED
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Queen Fabiola Children's University Hospital (Other)
Collaborators: Centre National de Référence S.aureus (Unknown)
Responsible Party: Sponsor
Other Study IDs: P2018/PNEUMO/PAPED
Record Dates: First submitted 2019-03-04; First posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-03

CONDITIONS: Cystic Fibrosis; Pseudomonas Aeruginosa; Cross Infection
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections; Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Respiratory secretions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cystic fibrosis patients with PA: All the children with acute or chronic Pseudomonas aeruginosa infection and followed-up in our cystic fibrosis center will be included in this study.

SUMMARY:
Cystic fibrosis is the most common hereditary autosomal recessive disease in the Caucasian population. The diseases is caused by a mutation of the gene coding for the CFTR protein (Cystic fibrosis transmembrane conductance regulator), an ion channel present at the apical pole of the epithelial cells. The channel dysfunction induces a deficit in hydration and a hyperviscosity of different exocrine secretions.

Clinically, Cystic fibrosis is a multi-systemic disease. Pulmonary and pancreatic involvement are classically in the foreground. Degradation of respiratory function, associated with acute and chronic infections, represents the major cause of morbidity and mortality.

Pseudomonas aeruginosa is a ubiquitous gram-negative bacillus found primarily in stagnant water. Pseudomonas aeruginosa is capable of colonizing the digestive, pulmonary and urinary mucosa and the skin. This bacterium is incriminated in many opportunistic infections including respiratory infections in patients with cystic fibrosis. Pseudomonas aeruginosa infection is the most common parenchymal lung infection in the Cystic fibrosis community.

Pseudomonas aeruginosa chronic carriage represents a factor of poor prognosis associated with an increase in morbidity and mortality. Complications related to chronic carriage of Pseudomonas aeruginosa justify the implementation of strategies of eviction, screening and eradication of acute Pseudomonas aeruginosa infection.

In addition to Pseudomonas aeruginosa contamination of patients via the environment, hand and airborne infections between patients with Cystic fibrosis have been reported. Measures to eliminate cross-transmissions have therefore been implemented in a majority of hospitals.

The aim of the study is firstly to identify the number of Pseudomonas aeruginosa cross-transmissions between patients with Cystic fibrosis followed-up in Cystic fibrosis center of HUDERF. Investigator will use the Pulsed-Field Gel Electrophoresis to assess the possibility of cross-infection.

Depending on the results, Investigator will implement new strategies to avoid future cross-contamination in our different places of care (consultation, hospitalization, physiotherapy…).

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis patients aged 0-20y followed in Cystic fibrosis at HUDERF
* For each participant, both parents or legally acceptable representative(s) must sign an informed consent form (ICF) indicating that they understand the purpose of, and procedures required for, the study and is willing to allow the child to participate in the study.
* Assent is also required of children capable of understanding the study (typically participants 7 years of age and older).

Exclusion Criteria:

* None

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cystic fibrosis patients followed-up in cystic fibrosis center in Brussels.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2019-02-06 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Identification of Pseudomonas cross infections between cystic fiborsis patients | through study completion
  Highlighting common strains (similar typing) of Pseudomonas aeruginosa in respiratory secretion using the PFGE (Pulsed-field Gel Electrophoresis)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe Beghin, MD, Principal Investigator — HUDERF
Locations (1):
- Hôpital Universitaire Des Enfants Reine Fabiola, Brussels, Belgium